CLINICAL TRIAL: NCT00576875
Title: Conte Centers for the Neuroscience of Depression
Brief Title: Duke Conte Center for the Neuroscience of Depression in Late Life
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00007678
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Major Depression
Keywords: Depression; Elderly; Neuroimaging; Postmortem; Knockout mouse
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood for DNA; Post-mortem brain tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Depressed: Older individuals with major depression
- Non-depressed: Older individuals without major depression

SUMMARY:
The proposed Silvio O. Conte Center for Neuroscience of Depression will focus on understanding the neurobiological mechanism of depression. A total of 5 projects are proposed. The center is focused on a single hypothesis. The first project examines localization of lesions, structural changes in critical regions subserving the circuit, alterations in the white matter tracts relevant to the circuit and changes in glutamate. The second project uses post mortem cell counting and cellular localization in serotonin receptors and assessment of the type of cell loss in the orbitofrontal cortex. The third project uses cognitive paradigms and functional MRI to probe the circuit and the role of brain lesions and serotonin on the functioning of this circuit. The fourth project uses transgenic and knockout mice to examine to role of norepinephrine and serotonin as it relates to the circuit. The final project is designed to assess in these transgenic mice using multielectrode array of single neuron recordings of the firing pattern of the circuit neurons in various states and tasks and the role of monoamines in modulating this circuit.

DETAILED DESCRIPTION:
Three shared resources, administrative, research and assessment and data management/statistics are proposed to facilitate the conduct of these projects and to ensure integration at the conceptual, analytical and resource availability level, and flow to the various projects. Findings from the center should greatly enhance our understanding of the biology of depressive disorders and help improve the treatment of these disorders. In addition, the technological innovations developed in the context of this project are likely to be of major importance and relevant to other studies of brain function.

ELIGIBILITY:
Inclusion Criteria:

For depressed group:

1. Age > 60 years
2. Major depression, single episode or recurrent
3. Ability to read and write English
4. MMSE >25
5. Willingness to participate in the follow-up study for at least two years.

For non-depressed group:

1. Age > 60 years
2. Ability to read and write English
3. MMSE >25
4. Willingness to participate in the follow-up study for at least two years

Exclusion Criteria:

1. Lifetime alcohol or drug dependence
2. Conditions associated with MRI abnormalities such hydrocephalus, benign and cancerous brain tumors, epilepsy, Parkinson's disease, Huntington's chorea, dementia, demyelinating diseases, etc.
3. Endocrine disorder (other than diabetes mellitus)
4. Any physical or intellectual disability that may affect completion of self rating instruments
5. Established clinical diagnosis of dementia
6. Other primary psychiatric disorders, including panic disorder, social phobia, OCD, non-affective psychosis (including schizo-affective disorder), schizophrenia, bipolar disorder
7. Any metal or pacemaker in the body which precludes MRI.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic; Outpatient psychiatry clinic; Inpatient psychiatry clinic; Self-referral
Sampling Method: Non-Probability Sample
Enrollment: 795 (Actual)
Dates: Start 2006-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Each of the projects in the Duke Conte Center has its own aims and primary outcomes | Up to five years

CONTACTS AND LOCATIONS:
Overall Officials: Ranga R Krishnan, MB, ChB, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States